CLINICAL TRIAL: NCT05412914
Title: The Impact of Remimazolam and Propofol on the Left Ventricular Systolic Performance During Anesthesia-induction for Non-cardiac Surgery: a Speckle Tracking Analysis of the Left Ventricular Strain Using Transthoracic Echocardiography
Brief Title: Remimazolam and Propofol on the Left Ventricular Strain During Anesthesia Induction for Non-cardiac Surgery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Konkuk University Medical Center (Other)
Responsible Party: Principal Investigator, Tae-Yop Kim, MD PhD, Professor, Department of Anesthesiology, Konkuk University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: 20210000-01
Record Dates: First submitted 2021-08-31; First posted 2022-06-09 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Surgical Procedure, Unspecified
MeSH Terms: interventions — Propofol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Remimazolam (Experimental): remimazolam infusion
  Interventions: Drug: Remimazolam infusion
- Propofol (Active Comparator): propofol infusion
  Interventions: Drug: Propofol infusion

INTERVENTIONS:
Drug: Remimazolam infusion — Remimazolam infusion for anesthesia induction
  Other Names: Byfavo
  Arms: Remimazolam
Drug: Propofol infusion — Propofol infusion for anesthesia induction
  Other Names: Fresofol
  Arms: Propofol

SUMMARY:
This study to compare the impacts of remimazolam or propofol on the left ventricular global longitudinal strain (LV-GLS) during anesthesia induction for non-cardiac surgery.

LV-GLS is analyzed by using speckle tracking technique of transthoracic echocardiography.

DETAILED DESCRIPTION:
This study to compare the impacts of remimazolam or propofol on the left ventricular global longitudinal strain (LV-GLS) during anesthesia induction for non-cardiac surgery (n=40).

Remimazolam or propofol is randomly administered for anesthesia induction (Group-R and Group-P, respectively) The changes of LV-GLS are analyzed by using using speckle tracking technique. For this study, 2-dimensional of transthoracic echocardiography LV images (apical 2-chamber, 3-chamber, and 4-chamber views) are recorded and stored before administration of remimazolam/propofol (T0), 2 minutes after the administration (T2), 4 minutes after the administration (T4), and 6 minutes after the administration (T6).

After the completion of the study, LV-GLS values at T0, T2, T4 and T6 are determined by the off-line analyses of the recorded and stored 2D-images.

For the off-line determination of LV-GLS, an automated software of speckle-tracking technique (Qapp Autostrain-LV™, Philips) is employed.

The primary measure:

Inter-group comparison of the lowest LV-GLS value out of LV-GLS values at T2, T4, and T6.

The secondary measures:

Inter-group comparisons of the LV-GLS values at T0, T2, T4 and T8. Intra-group comparisons of the LV-GLS value at T0 vs. those at T2, T4 and T8

ELIGIBILITY:
Inclusion Criteria:

* left ventricular ejection fraction> 50%
* no left ventricular regional wall motion abnormality

Exclusion Criteria:

* atrial fibrillation
* unfavorable airway
* hypotension requiring inotropic support

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-01-26 (Actual); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
the averaged longitudinal strain of the left ventricle (%) | 2.5 minutes
  inter-group comparisons of the lowest values of the longitudinal strains of the left ventricle in the transthoracic echocardiography after administering remimazolam- or propofol-administration for anesthesia induction

SECONDARY OUTCOMES:
the longitudinal strain of the left ventricle in apical long-axis view (%) | 2.5 minutes
  inter-group comparisons of the longitudinal strains of the left ventricle in apical long-xis view of the transthoracic echocardiography after administering remimazolam- or propofol-administration for anesthesia induction
the longitudinal strain of the left ventricle in apical 2 chamber view (%) | 2.5 minutes
  inter-group comparisons of the longitudinal strains of the left ventricle in apical 2 chamber view of the transthoracic echocardiography after administering remimazolam- or propofol-administration for anesthesia induction
the longitudinal strain of the left ventricle in apical 4 chamber view (%) | 2.5 minutes
  inter-group comparisons of the longitudinal strains of the left ventricle in apical 4 chamber view of the transthoracic echocardiography after administering remimazolam- or propofol-administration for anesthesia induction
the election fraction of the left ventricle | 2.5 minutes
  inter-group comparisons of the ejection fraction of the left ventricle in the transthoracic echocardiography after administering remimazolam- or propofol-administration for anesthesia induction

CONTACTS AND LOCATIONS:
Overall Officials: Tae-Yop Kim, MD, PhD, Principal Investigator — Konkuk University Medical Center
Locations (1):
- Konkuk University Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No